CLINICAL TRIAL: NCT01130558
Title: Efficacy of Structured Insulin Orders in Improving Glycemic Control
Brief Title: Efficacy of Structured Insulin Order
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Enrico Cagliero, M.D., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008P-0022131
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; basal-bolus insulin; insulin ordering
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ordering template and education (Active Comparator): Internal medical residents who were asked to use the insulin order template and received education about basal-bolus insulin ordering.
  Interventions: Other: Diabetes Management
- Education (Active Comparator): Internal medical residents who received education about basal-bolus insulin ordering.
  Interventions: Other: Diabetes Management

INTERVENTIONS:
Other: Diabetes Management — Using electronic insulin order template for basal-bolus insulin and education

SUMMARY:
The purpose of this study is to determine whether an electronic order template for basal-bolus insulin will improve mean blood glucose in hospitalized general medical patients with poorly controlled type 2 diabetes.

DETAILED DESCRIPTION:
The study randomly assigned internal medicine residents to use an electronic insulin order template plus basal-bolus ordering education versus education only. For all patients with uncontrolled type 2 diabetes treated by these physicians, mean blood glucose, rate of hypoglycemia, and rate of sliding scale insulin use were measured.

ELIGIBILITY:
Inclusion Criteria:

* Blood glucose less than 60 mg/dl or greater than 180 mg/dl during hospital stay

Exclusion Criteria:

* Diagnosis of Type 1 Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Mean blood Glucose | 6 days

SECONDARY OUTCOMES:
rates of glucose values less than 60 mg/dl or less than 40 mg/dl | 6 days
rate of use of sliding scale insulin | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Cagliero, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States